CLINICAL TRIAL: NCT02251093
Title: Study of the Efficacy and Tolerance of Intra-vaginal Treatment With a Total Freeze-dried Culture of Lcr Regenerans® in the Prevention of Relapses of Recurrent Vulvovaginal Candidiasis. International Phase III, Randomised, Multi-centre, Parallel-group, Two Arm, Double-blind Superiority Trial Versus Placebo.
Brief Title: Study of the Efficacy and Tolerance of Intra-vaginal Treatment With a Total Freeze-dried Culture of Lcr Regenerans® in the Prevention of Relapses of Recurrent Vulvovaginal Candidiasis
Acronym: GYNOCANS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Probionov (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO_2013 - 02; 2013-002480-26 (EudraCT Number)
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Candidiasis, Vulvovaginal
Keywords: mycosis; vulvovaginal candidiasis; lcr35; Lcr Regenerans®
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Mycoses

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lcr Regenerans (Experimental)
  Interventions: Drug: Lcr Regenerans
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lcr Regenerans — Dosage: 1 vaginal capsule per day Route of administration: intravaginal Treatment duration: One 21-day cycle
  Other Names: GYNOPHILUS
  Arms: Lcr Regenerans
Drug: Placebo — Dosage: 1 vaginal capsule per day Route of administration: intravaginal Treatment duration: One 21-day cycle
  Arms: Placebo

SUMMARY:
The trial medicinal product (Lcr Regenerans®) is obtained from the culture of a strain of Lactobacillus rhamnosus Lcr35®. By virtue of the freeze-drying technique, Lactobacillus rhamnosus Lcr35® is a live bacterium administered with its culture medium.

It should be noted that Lcr Regenerans® is already marketed as a medical device (EC marking: 0499). It helps to regenerate the vaginal flora thanks to its physical and chemical effects (lowering the vaginal pH).

A number of in vitro and in vivo studies have demonstrated the ability of Lactobacillus rhamnosus Lcr35®:

* to establish itself in the vaginal epithelium, along with the durability of this establishment.
* and to inhibit the growth of pathogenic organisms responsible for causing bacterial vaginosis (Gardnerella vaginalis and Prevotella bivia) but also for mycoses (Candida albicans), by synthesising various microbicidal substances.

This research follows on from the Candiflore observational study in which 514 patients were monitored and which demonstrated a clearly positive result in favour of the use of vaginal Lcr Regenerans® for preventing recurrences of VVC.

The purpose of this new research is thus to demonstrate the efficacy of Lcr Regenerans®, in the prevention of vulvovaginal candidiasis recurrences in patients with a history of VVC with recurrent episodes, in view of obtaining a marketing authorisation.

DETAILED DESCRIPTION:
Treatment of RVVC is difficult due to the multi-factor nature of recurrences and of the poorly understood local immune dysfunctions that may arise. The oral or topical antifungal maintenance treatment usually recommended is for a period of 6 months, though the VVC relapse rate is high, with 60 to 70% of women presenting with a recurrence within 2 months following termination of treatment. Moreover, antifungal agent-related adverse events are frequent and their long-term use can be conducive to the onset of bacterial vaginosis (BV).

The vaginal administration of probiotic strains (Lactobacillus) capable of regenerating the vaginal flora and of inhibiting the development of Candida albicans and/or its adhesion to the vaginal epithelium, would appear to be an interesting therapeutic alternative for preventing VVC recurrences.

The trial medicinal product (Lcr Regenerans®) is obtained from the culture of a strain of Lactobacillus rhamnosus Lcr35®. By virtue of the freeze-drying technique, Lactobacillus rhamnosus Lcr35® is a live bacterium administered with its culture medium.

It should be noted that Lcr Regenerans® is already marketed as a medical device (EC marking: 0499). It helps to regenerate the vaginal flora thanks to its physical and chemical effects (lowering the vaginal pH).

A number of in vitro and in vivo studies have demonstrated the ability of Lactobacillus rhamnosus Lcr35®:

* to establish itself in the vaginal epithelium, along with the durability of this establishment.
* and to inhibit the growth of pathogenic organisms responsible for causing bacterial vaginosis (Gardnerella vaginalis and Prevotella bivia) but also for mycoses (Candida albicans), by synthesising various microbicidal substances.

This research follows on from the Candiflore observational study in which 514 patients were monitored and which demonstrated a clearly positive result in favour of the use of vaginal Lcr Regenerans® for preventing recurrences of VVC.

The purpose of this new research is thus to demonstrate the efficacy of Lcr Regenerans®, in the prevention of vulvovaginal candidiasis recurrences in patients with a history of VVC with recurrent episodes, in view of obtaining a marketing authorisation.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from recurrent VVC (RVVC) defined by the existence of at least 4 VVC episodes during the past year, including the one concerned by the screening visit In addition to the current episode, at least one episode occurring during the two previous years must also have been documented by mycological examination
* Patient suffering from acute vulvovaginitis characterised by the presence of the following clinical criteria at V1 (pruritus symptoms, vulvovaginal signs such as erythema, vaginal discharge)
* Patient with a positive mycological examination at V1
* Patient cured in clinical terms 8 days after treatment with MONAZOL 300 mg vaginal suppositories (one suppository at night before sleep, single administration) and followed by the application of MONAZOL 2 pourcent cream (8-day treatment)
* Woman of child-bearing age with a negative urine pregnancy test and using a means of contraception deemed effective by the investigator (excluding spermicides) throughout the trial
* Patient/Legal representative able to speak and read the local language, having been informed of the trial and having voluntarily signed an Informed Consent Form
* Patient/Legal representative registered with a social insurance scheme

Exclusion Criteria:

* Presence of a presumed or proven, gynaecologically-related bacterial or viral infection, whether treated or not during the month preceding the inclusion, or present at the time of inclusion.
* Presence of an existing gynaecological infection that could interfere with the assessment of the trial treatment (severe cervical dysplasia or carcinoma in situ, invasive carcinoma, intra-epithelial cervical neoplasia, squamous intra-epithelial lesions etc.)
* Patients with a negative mycological examination at V1
* Lack of adequately documented previous episodes to assert the recurrent nature of the VVC (4 episodes in one year, two of which documented by mycological examination over the past two years [thus, in addition to the current episode, at least one episode occurring during the two previous years must also have been documented by mycological examination])
* Antifungals taken by general route (in particular Fluconazole) during the month preceding the screening visit, in view of preventing recurrences (the treatment of an acute VVC episode is not an exclusion criterion).
* Use of probiotics in the month preceding the screening visit.
* Use of prebiotics (acidifiers) during the two weeks preceding the screening visit.
* Allergy to one of the active ingredients or one of the excipients in the products.
* Patient unable to comply with the constraints of the Protocol.
* Breastfeeding patient.
* Patient with menstrual bleeding lasting more than 8 days a month.
* Post-menopausal women with last menstrual period at least 12 months prior to screening
* Patient having taken part in a clinical trial in the 3 months preceding inclusion in the present Protocol.
* Patient with a severe acute or chronic disease deemed by the Investigator to be incompatible with participation in the trial, or a serious infection that is life-threatening in the short term.
* Immuno-suppressed patient.
* Patient presenting with a previous illness which, according to the Investigator, is likely to interfere with the results of the trial or expose the patient to an additional risk.
* Patient linguistically (unable to speak or write the local language) or mentally unable to understand and sign the Informed Consent Form.
* Patient deprived of her liberty by order of the Courts or civil authorities or subject to a guardianship order.
* Patient likely not to comply with treatment.
* Patient unable to be contacted in the case of an emergency.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2014-05; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Recurrence confirmed by a mycological test, occurring during the treatment period, or within 5 months of trial treatment termination | 5 months
  The main outcome measure chosen for this trial is the rate of clinical recurrence confirmed by a mycological test, occurring during the treatment period, or within 5 months of trial treatment termination (fraction of patients presenting with at least one recurrence during the treatment period or during the 5-month monitoring period).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe JUDLIN, Principal Investigator — Maternité Régionale Universitaire de Nancy
Locations (1):
- Probionov, Aurillac, France